CLINICAL TRIAL: NCT04772001
Title: Clinical Study of Hydrochloride Anlotinib Combined With Concurrent Radiochemotherapy for Locally Advanced (Stage IB3 and IIA2-IVA) Cervical Cancer
Brief Title: Concurrent Radiochemotherapy Plus Anlotinib for Locally Advanced Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Hui Qiu, Chief Physician and Director of Department of Radiation and Medical Oncology (Gynaecologic Oncology, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-RT-ALTER-01
Record Dates: First submitted 2021-02-19; First posted 2021-02-25 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Uterine Cervical Neoplasms; Chemoradiotherapy; Angiogenesis
Keywords: Uterine Cervical Neoplasms; Chemoradiotherapy; Anlotinib
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Carboplatin; Brachytherapy

STUDY DESIGN:
Intervention Model Description: All participants will be included in one arm and receive chemoradiotherapy and anlotinib according to the protocol
Masking Description: No mask.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCRT+Anlotinib (Experimental): Classical chemoradiotherapy will be conducted by clinical routine method. Radiation will be given by external beam of 45Gy total dose and 3D-brachytherapy of 30Gy/5F or 28Gy/4F. Duration of radiotherapy will be no more than 8 weeks. Concurrent chemotherapy will be administrated weekly during radiation for a total of 5-6 doses. Cisplatin of 40mg/m2 will be the most preferred regime and for patients with intolerable toxicity of cisplatin, carboplatin of AUC 2 will be the alternative drug. Hydrochloride anlotinib will be orally taken daily at a dose level of 12mg for 14 days. Then rest for 7 days and start a new cycles for a total of 3 cycles. First capsule of anlotinib will be taken 7 days before the first radiation.
  Interventions: Drug: Hydrochloride anlotinib; Drug: cis Platinum/carboplatin; Radiation: External beam radiotherapy and brachytherapy

INTERVENTIONS:
Drug: Hydrochloride anlotinib — Hydrochloride anlotinib is a small molecular anti-angiogenesis drug with multiple targets. It will be taken at a starting dose of 12 mg for 14 days. Then participants will rest for 7 days and start a new cycles. At most of 3 cycles will be administrated. If intolerable toxicity happen, dosage of 10mg or 8mg will be taken.
Drug: cis Platinum/carboplatin — Concurrent chemotherapy will be administrated weekly during radiation for a total of 5-6 doses. Cisplatin of 40mg/m2 will be the most preferred regime. For patients with intolerable toxicity of cisplatin, carboplatin of AUC 2 will be the alternative drug.
Radiation: External beam radiotherapy and brachytherapy — Radiation will be given by external beam of 45Gy total dose and 3D-brachytherapy of 30Gy/5F or 28Gy/4F. Duration of radiotherapy will be no more than 8 weeks.

SUMMARY:
To observe the efficacy and safety of hydrochloride anlotinib combined with concurrent radiochemotherapy for patients with FIGO stage IB3 and IIA2-IVA cervical cancer. Patient characteristics, image and genetic information of tumor, microbial sample of tumor microenvironment and biomarker in the blood sample will be collected and analysis by multi-omics and bioinformatic technology. Aim to provide a new treatment module for cervical cancer.

DETAILED DESCRIPTION:
Patients diagnosed pathologically as cervical cancer (squamous carcinoma, adenocarcinoma or adenosquamous carcinoma) with stage of FIGO IB3 and IIA2 to IVB will be included in this study according to the prescribed criteria in the protocal. Classical radiochemotherapy will be conducted by clinical routine method. Radiation will be given by external beam radiation of 45Gy total dose and 3D-brachytherapy of 30Gy/5F or 28Gy/4F. Duration of radiotherapy will be no more than 8 weeks. Concurrent chemotherapy will be administrated weekly during radiation for a total of 5-6 doses. Cisplatin of 40mg/m2 will be the most preferred regime and for patients with intolerable toxicity of cisplatin, carboplatin of AUC 2 will be the alternative drug. Apart from that, hydrochloride anlotinib, a multiple targets anti-angiogenesis kinase approved by CFDA, will be orally taken daily at a dose of 12mg for 14 days aiming to improve tumor response. Then rest for 7 days and start a new cycles for a total of 3 cycles. First capsule of anlotinib will be taken 7 days before the first radiation. Once the treatment is finished, patients will be examination for tumor evaluation and toxicity monitor every 3 months for the first 2 years and then every half years for the third year unless progression or death. During those period, patient characteristics, image data, tumor tissue, blood, urine, stool and microbial sample of tumor micro environment will be collected and analysis by multi-omics and bioinformatic technology. A total of 53 patients will be included and this study will be conducted in the department of radiation and clinical oncology in Zhongnan Hospital of Wuhan University.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old;
2. ECOG PS score 0-2 points;
3. After pathological examination, it is clear that it is cervical cancer, the pathological types include squamous cell carcinoma, adenocarcinoma and adenosquamous carcinoma;
4. The staging conforms to the definitions of IB3 and IIA2-IVA in FIGO2018;
5. The expected survival period is ≥6 months;
6. The lesion meets the requirements of RECIST 1.1 for evaluable lesions;
7. Have not received any form of anti-tumor treatment before joining the group (except for partial cervical biopsy resection);
8. Expect to tolerate radiotherapy;
9. It is expected to tolerate concurrent chemotherapy with platinum drugs;
10. It is expected to tolerate oral Anlotinib treatment;
11. The sitting blood pressure at rest is less than the normal high value (<140/90mmHg), or the average blood pressure of the 24-hour ambulatory blood pressure monitoring is less than the normal high value (<140/90mmHg), regardless of whether you are taking antihypertensive drugs or not;
12. Hematology indicators meet (no blood transfusion and no correction with hematopoietic stimulating factor drugs within 7 days before screening): white blood cell count (WBC) ≥3.5×109/L and ≤10×109/L, neutrophil count ( ANC) ≥1.5×109/L, platelet (PLT) ≥125×109/L, hemoglobin (Hb) ≥90g/L;
13. The liver function index meets: ALT and AST≤2.5 times high normal value (ULN), bilirubin≤1.5×ULN, albumin≥35g/L;
14. The coagulation function index meets (not receiving anticoagulation or drug hemostasis treatment): PT and APTT ≤ 1.5×ULN, and INR ≤ 1.5 ULN;
15. Renal function indicators meet: urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN and creatinine clearance ≥60 mL/min (Cockcroft-Gault formula), urine protein <2+ or 24-hour urine protein quantitative <1g
16. Women of childbearing age must undergo a serum pregnancy study within 7 days before the first medication, and the result is negative, and they are not breastfeeding. Female subjects of childbearing age must agree to use effective methods of contraception during the study period and within 180 days after the last administration of the study drug;
17. Obtain informed consent signed by the patient or his legal representative;
18. Have good compliance.

Exclusion Criteria:

1. Any unstable systemic disease, including but not limited to active infection within 4 weeks (defined as fever with a body temperature exceeding 38.5℃ or clear evidence of bacteremia or evidence of heart, brain, kidney, lung, etc.) Infectious changes in the liver and intestines), circulatory accidents within 6 months (malignant hypertension, myocardial infarction, severe/unstable angina pectoris, heart insufficiency above NYHA level 2, clinically significant supraventricular or Ventricular arrhythmia, cerebrovascular accident that has not recovered or caused serious sequelae), uncontrolled type 2 diabetes (fasting blood glucose> 11.1mmol/L or glycosylated hemoglobin> 8%), lung insufficiency (pulmonary function caused by any reason Decrease, defined as lung function test FEV1/FVC<70%, FEV1<80% predicted value).
2. Past autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, autoimmune liver disease, autoimmune thyroiditis, systemic vasculitis, scleroderma, dermatomyositis, self Immune hemolytic anemia;
3. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; hepatitis C, defined as HCV -RNA is higher than the detection limit of the analysis method) or combined with hepatitis B and C infection;
4. The history of live attenuated vaccine vaccination within 28 days before the first study medication or the expected live attenuated vaccine vaccination during the study period;
5. Imaging shows that the tumor invades large blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the follow-up study or other diseases with serious bleeding risk (the bleeding caused by simple cervical tumor rupture is not included)
6. Previously received anti-angiogenesis targeted drug therapy, or other treatments for VEGFR inhibitors;
7. There is evidence of active tuberculosis infection within 1 year before screening;
8. Any other malignant tumor has been diagnosed within 5 years before entering the study, except for fully treated basal cell carcinoma or squamous cell skin cancer or cervical carcinoma in situ;
9. Major surgery has been performed within 28 days before randomization (tissue biopsy required for diagnosis and central venous catheter insertion via peripheral venipuncture [PICC] are allowed);
10. Arteriovenous thrombosis events that occurred within 6 months before randomization, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis (venous thrombosis caused by intravenous catheterization due to pre-chemotherapy, which has been cured by the investigator Except) and pulmonary embolism;
11. Subjects who have previously received or plan to receive allogeneic bone marrow transplantation or solid organ transplantation;
12. There is intestinal obstruction with significant clinical significance, intestinal repair, intestinal anastomosis or intestinal fistula occurs at any time for any reason;
13. Subjects with symptoms of hemoptysis and the maximum daily volume of hemoptysis ≥2.5 mL within 2 months before entering the study. Have had significant clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months before entering the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline stool occult blood++ or above, or suffering from vasculitis, etc.; Known to have inherited or acquired bleeding and thrombotic tendency, such as: hemophilia, blood coagulation disorder, thrombocytopenia, hypersplenism, etc.;
14. Macroscopic hematuria or urinary bleeding indicated by other evidence;
15. Are receiving thrombolysis or need long-term anticoagulation therapy with warfarin or heparin, or need long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day)
16. Peripheral neuropathy ≥ Grade 2;
17. Intolerance to platinum chemotherapy drugs (including intolerance caused by allergies or other physical symptoms);
18. Kidney stones at risk of seizure, one kidney has no function or anatomically single kidney;
19. Long-term bed rest for any reason;
20. Cachexia state;
21. Known allergy to Anlotinib or any of its excipients;
22. Those who have other anti-tumor treatment plan during treatment;
23. Participated in any other drug clinical research within 4 weeks before randomization, or no more than 5 half-lives from the last study drug;
24. The subject is known to have a history of psychotropic drug abuse, alcohol abuse or drug abuse;
25. Those who have a mental illness that seriously affects cognition and cannot achieve a stable mental state;
26. According to the judgment of the investigator, the patient may have other factors that may cause the study to be terminated halfway, such as other serious diseases or severe laboratory abnormalities or other factors that will affect the safety of the subjects, or test data And the family or society where the sample was collected

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
3 years disease free survival rate | 3 years from enrollment
  Proportion of participants without tumor recurrence or death at 3 years from enrollment

SECONDARY OUTCOMES:
Adverse events | From enrollment to 90 days after treatment finish
  Adverse events data according to CTCAE version 5.0
3 years overall survival rate | 3 years from enrollment
  Proportion of survival participants at 3 years from enrollment
Objective response rate | 5 years from enrollment
  Proportion of participants with complete response and partial response
Disease control rate | 5 years from enrollment
  Proportion of participants with complete response, partial response and stable disease
5 years progression free survival rate | 5 years from enrollment
  Proportion of participants without tumor progression or death at 3 years from enrollment
5 years overall survival rate | 5 years from enrollment
  Proportion of survival participants at 5 years from enrollment
Median overall survival | 5 years of follow-up
  Median survival time of all participants from enrollment to death of any reason
Median progression free survival | 5 years of follow-up
  Median time of all participants from enrollment to tumor progression
Score of life quality | 3 years from enrollment
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire. Scores ranging from 0 to 100, higher scores indicating better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Qiu, Ph. D., Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krill LS, Tewari KS. Integration of bevacizumab with chemotherapy doublets for advanced cervical cancer. Expert Opin Pharmacother. 2015 Apr;16(5):675-83. doi: 10.1517/14656566.2015.1010511. Epub 2015 Feb 3. PMID 25643984
- [Background] Monk BJ, Sill MW, Burger RA, Gray HJ, Buekers TE, Roman LD. Phase II trial of bevacizumab in the treatment of persistent or recurrent squamous cell carcinoma of the cervix: a gynecologic oncology group study. J Clin Oncol. 2009 Mar 1;27(7):1069-74. doi: 10.1200/JCO.2008.18.9043. Epub 2009 Jan 12. PMID 19139430
- [Background] Schefter T, Winter K, Kwon JS, Stuhr K, Balaraj K, Yaremko BP, Small W Jr, Sause W, Gaffney D; Radiation Therapy Oncology Group (RTOG). RTOG 0417: efficacy of bevacizumab in combination with definitive radiation therapy and cisplatin chemotherapy in untreated patients with locally advanced cervical carcinoma. Int J Radiat Oncol Biol Phys. 2014 Jan 1;88(1):101-5. doi: 10.1016/j.ijrobp.2013.10.022. PMID 24331655
- [Background] Youn SH, Kim YJ, Seo SS, Kang S, Lim MC, Chang HK, Park SY, Kim JY. Effect of addition of bevacizumab to chemoradiotherapy in newly diagnosed stage IVB cervical cancer: a single institution experience in Korea. Int J Gynecol Cancer. 2020 Jun;30(6):764-771. doi: 10.1136/ijgc-2020-001200. Epub 2020 Apr 9. PMID 32276937
- [Background] Han B, Li K, Zhao Y, Li B, Cheng Y, Zhou J, Lu Y, Shi Y, Wang Z, Jiang L, Luo Y, Zhang Y, Huang C, Li Q, Wu G. Anlotinib as a third-line therapy in patients with refractory advanced non-small-cell lung cancer: a multicentre, randomised phase II trial (ALTER0302). Br J Cancer. 2018 Mar 6;118(5):654-661. doi: 10.1038/bjc.2017.478. Epub 2018 Feb 13. PMID 29438373